CLINICAL TRIAL: NCT03418753
Title: Non-invasive Diagnostic for Assessing Elevated Intracranial Pressure
Status: Completed | Type: Observational
Sponsor: Oculogica, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ICP001
Record Dates: First submitted 2018-01-17; First posted 2018-02-01 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Intracranial Pressure Increase
Keywords: noninvasive diagnosis
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- single: subjects with abnormal intracranial pressure
  Interventions: Diagnostic Test: EyeBOX for ICP

INTERVENTIONS:
Diagnostic Test: EyeBOX for ICP — non-invasive ICP Score algorithm using eye-tracking data from the EyeBOX(TM) device, which tracks the movement of the pupils over time

SUMMARY:
The study is a prospective, multi-center, non-randomized, open label observational study. The objective of this study is to compare the accuracy of the EyeBOX to a clinical diagnosis of abnormal ICP as determined by an external ventriculostomy drain (EVD) or ventriculostomy catheter.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. Require placement of an ICP monitor or ventriculostomy catheter for clinical purposes.
3. Be between the ages of 4 and 70 years old.
4. Have baseline vision correctable to within 20/500 bilaterally.
5. Have no prior history of ocular dysmotility.
6. Be awake with spontaneous eye opening at the time when eye tracking is performed.

Exclusion Criteria:

1. Have a prior history of strabismus, diplopia, or palsy of CN-III, IV or VI.
2. Be blind (no light perception), have missing eyes, be unable to open their eyes.
3. Have a prior history of ocular motility dysfunction.
4. Have had extensive prior eye surgery.
5. Have any physical or mental injury or baseline disability rendering task completion difficult.
6. Be intoxicated or have blood alcohol level greater than 0.2.
7. Be a prisoner or in the company of a police officer or law enforcement officer pending arrest.

Ages: 4 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study will enroll pediatric and adult patients with abnormal ICP. Subjects who meet all of the inclusion criteria and none of the exclusion criteria will be considered for enrollment into the study. There will be no enrollment restrictions based on race, ethnic origin, gender, or pregnancy status and efforts will be made to ensure that the benefits and burdens of research participation are distributed in an equitable manner. Subjects must require ICP monitoring for clinical indications. At the time when eye tracking is performed all patients must be awake with spontaneous eye opening.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity | from time of enrollment through the period that ICP monitoring is required for clinical purposes up to 104 weeks
  EyeBOX assessment of abnormal ICP relative to invasive intracranial pressure monitor

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jackson, MD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kolecki R, Dammavalam V, Bin Zahid A, Hubbard M, Choudhry O, Reyes M, Han B, Wang T, Papas PV, Adem A, North E, Gilbertson DT, Kondziolka D, Huang JH, Huang PP, Samadani U. Elevated intracranial pressure and reversible eye-tracking changes detected while viewing a film clip. J Neurosurg. 2018 Mar;128(3):811-818. doi: 10.3171/2016.12.JNS161265. Epub 2017 Jun 2. PMID 28574312